CLINICAL TRIAL: NCT06378099
Title: Evaluation of the Effect of Consensus-based Protocols for the Treatment of Minor Ailments in Drugstores and Pharmacies in Medellin and the Metropolitan Area, Colombia: A Randomized Clinical Trial.
Brief Title: Evaluation of the Effect of Consensus-based Protocols for the Treatment of Minor Ailments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Farmacias Pasteur (Unknown)
Responsible Party: Principal Investigator, Pedro Amariles, Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CBP Colombia
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Community Pharmacy Services
Keywords: Minor ailments; Minor Ailment Services; Pharmacies; Nonprescription drugs; Pharmacy Technicians; Health education; Self care; Ambulatory care; Community Health Services
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: An exploratory, clustered randomized controlled clinical trial with a baseline period will be conducted over a 10-month period. During this time, five MA will be analyzed: influenza-like syndrome and catarrh, headache, common cold, sore throat, and menstrual pain or cramps. Drugstores and pharmacies (clusters) will be randomized in a 1:1 ratio to either the intervention group (management using CBPs) or the control group (standard management + education on responsible self-medication).
Masking Description: Blinding of the participants and the pharmacists involved in the care is not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (standard management + education on responsible self-medication) (No Intervention): Patients will receive standard management + education on responsible self-medication. This group will have three activities: 1. Voluntary selection of OTC medication, 2. Health education on what responsible self-medication entails, 3. Monitoring for moderate and serious ADRs related to the use of selected nonprescription drugs or worsening symptoms of the MA, with referral to a GP if necessary.
  For each MA, the Pharmacist will request the patient's signature on Annex 1, proceed with Activity 1, fill in the instrument included in Annex 4, and continue with Activity 2.
  On days 3, 5, 7, and 10 after the consultation, patients will be contacted via a chatbot or a phone call to answer Annex 5. On days 5 to 6, and 10 to 12, a pharmacist of the research team will review patient responses to evaluate the need for medical referral (Activity 3), if the presence of a moderate or serious ADR or worsening of the symptom is identified (T5-T6, T10-T12).
- Intervention Group (management using CBPs) (Experimental): Patients will receive management using CBPs. This group will have four activities: 1. Identification and classification of the MA, 2.Referral to a GP if the patient's condition is not classified as an MA, 3. Patient guidance on appropriate pharmacological measures in case an OTC medication is required 4. Monitoring for moderate or serious ADRs related to the use of selected nonprescription drugs or worsening symptoms of the MA, with referral to a GP if necessary.
  For each MA, the Pharmacist will request the patient's Informed Consent, apply what is described in Activities 1, 2, and 3, and fill in the instrument included in Annex 4.
  Days 3, 5, 6, 7, 10, and 12 will be followed as described for control group.
  Interventions: Other: Patient guided and followed by the pharmacist

INTERVENTIONS:
Other: Patient guided and followed by the pharmacist — The Study Coordinating Group will train the pharmacy Staff regarding these protocols.
  This training will cover both pharmacological and non-pharmacological aspects of MA management. The pharmacological component will emphasize the appropriate selection and safe use of nonprescription drugs, with a focus on identifying potential drug interactions, contraindications, and moderate and serious ADRs. Pharmacy staff will also be equipped with tools to apply proper criteria for referral to a GP when necessary.
  The staff will be divided into three groups, and every group will have a minimum of two sessions, each one of 4 hours. Additionally, there will be a practical component where simulations of real situations will be conducted.
  Throughout the 12-month follow-up and intervention period, one of the researchers will be available to receive phone calls to address doubts and concerns about the Consensus-based Protocols.
  Other Names: Use of consensus-based protocols
  Arms: Intervention Group (management using CBPs)

SUMMARY:
Minor ailments are common, self-limited conditions unrelated to the patient's underlying health problems or adverse effects of their current medications. Minor ailment services are pharmacist-led interventions that provide patients with the most appropriate recommendation when unsure about the medication for a specific minor ailment. It involves advice on nonprescription drugs, non-pharmacological measures, or referral to another health care practitioner. In Colombia, evaluating and implementing this service could optimize nonprescription drugs use and improve minor ailment management in primary health care settings.

DETAILED DESCRIPTION:
A 10-month parallel-group clinical trial will be conducted in drugstores and pharmacies (ambulatory retail establishments) in Medellín and the Metropolitan Area. Patients requesting nonprescription drugs for one of five predefined minor ailments (influenza-like syndrome, common cold, headache, dysmenorrhea, or sore throat) will be eligible. Establishments, randomized by cluster sampling, will be allocated to either the intervention (management using CBPs) or control (standard management + education on responsible self-medication) group. Pharmacy staff will receive training in appropriate CBP use. Eligible patients will be consecutively enrolled and followed-up by the research team on days 3, 5, 7, and 10 after the consultation in both groups. Analyses will be performed using Python, including descriptive statistics, bivariate comparisons (p < 0.05), and multivariate Cox regression for significant variables. An intention-to-treat approach will address missing data and dropouts.

The aim of this study is to evaluate the effect of Consensus-based Protocols (CBPs) on the management and duration of some MA, and on the referral rate to General medical Practitioner (GPs) in drugstores and pharmacies. Secondary outcomes include: 1) To clinically and socio-demographically characterize the population that visits a drugstore or pharmacy requesting a nonprescription drug to manage a MA, and 2) To assess the management, duration, rate and causes of GP referrals in drugstores and pharmacies with the use of CBPs among patients requesting nonprescription drugs for the management of a potential MA.

ELIGIBILITY:
Inclusion Criteria:

Drugstores and drugstores/pharmacies:

* Establishments located in Medellin and Metropolitan area
* Establishments that have a Pharmacy Technician serving as the technical director.
* Establishments with electronic point-of-sale system for data collection.
* Commitment to participate for the full 10-month study period.

Participants (patients):

* Explicit consent to participate in the study.
* Are the direct consumers requesting the nonprescription drug (i.e., not requesting them on behalf of someone else).
* Present one of the five predefined potential MA that will be included in the study: influenza-like syndrome and catarrh, headache, common cold, sore throat, and menstrual pain or cramps.
* Have access to mobile phone for follow-upThe person requesting the OTC medication must be the end consumer of it.

Exclusion Criteria:

* Subjects who refuse to sign the informed consent
* Subjects with an evident incapacity to complete the data questionnaire
* Pregnant or breastfeeding women
* Patients whose MA result from an ADR
* Patients with symptoms lasting more than seven days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
MA resolution | 12 months
  MA resolution will be evaluated using five self-administered questionnaires. These will be administered at baseline (T0) before the intervention, and on days 3 (T3), 5 (T5), 7 (T7), and 10 (T10) after the consultation.
  MA resolution will be recorded as a binary outcome (yes/no). This outcome is clinically relevant as it will reflect the effectiveness of the intervention with CBPs.
MA duration | 12 months
  The duration of the MA will be evaluated using five self-administered questionnaires. These will be administered at baseline (T0) before the intervention, and on days 3 (T3), 5 (T5), 7 (T7), and 10 (T10) after the consultation.
  MA duration will be measured in days from the intervention at the drugstore or pharmacy to complete symptom resolution or if a referral to a GP is needed. This outcome is clinically relevant as it will reflect the effectiveness of the intervention with CBPs.
Referral rate to GP | 12 months
  Referral rate to GP, both due to symptoms worsening or occurrence of moderate or serious ADRs, will be evaluated using five self-administered questionnaires. These will be administered at baseline (T0) before the intervention, and on days 3 (T3), 5 (T5), 7 (T7), and 10 (T10) after the consultation.
  Based on patients' responses to follow-up questionnaires, referral to a GP will be recorded as a binary outcome (yes/no), indicating whether a referral occurred due to symptom worsening or suspected moderate or serious ADRs. This measure is relevant for evaluating patient safety and the effectiveness of the intervention with CBPs.

SECONDARY OUTCOMES:
Characterization of the patient population visiting the drugstores and pharmacies to request nonprescription drugs for the management of a MA | 3 months
  Sociodemographic and clinical data (e.g., age, sex, education level, prior use of nonprescription drugs) will be collected only at baseline (T0), before the intervention. This data will help contextualize the findings and identify population-specific factors influencing outcomes.
Identification and classification of the MA | 12 months
  In both the intervention and control groups, the presence and type of MA will be recorded at baseline (T0). In the control group (standard management + education on responsible self-medication), the patient will self-identify and classify the MA, whereas in the intervention group (management using CBPs), this will be done by the pharmacy staff following protocolized classification criteria. The outcome is relevant to verify the presence of a MA within drugstores and pharmacies.
Need for a nonprescription drug to treat the MA | 12 months
  This binary variable (yes/no) will be assessed in both groups at baseline (T0) and will indicate whether the patient obtained a nonprescription drug for MA management. In the control group (standard management + education on responsible self-medication), medication selection will be driven by the patient's decision. In the intervention group (management using CBPs), this decision will be guided by the pharmacy staff in accordance with the CBPs. Clinically, this informs the appropriateness and potential rationalization of nonprescription drug use under protocol-based pharmaceutical guidance.

CONTACTS AND LOCATIONS:
Locations (1):
- Farmacias Pasteur S.A., Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
Confidentiality of information will be assured, ensuring that the collected data remains anonymous and will not be disclosed at any phase of the trial (results, publications, or result presentations).